CLINICAL TRIAL: NCT03092583
Title: Analysis of DNA Methylation in Spondyloarthritis
Acronym: METYLAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P/2015/252
Record Dates: First submitted 2017-03-17; First posted 2017-03-28 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Spondylitis, Ankylosing; Axial Spondyloarthritis; DNA Methylation
MeSH Terms: conditions — Spondylitis, Ankylosing; Axial Spondyloarthritis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group (Experimental): Subjects must meet the modified New York criteria for AS, or the ASAS criteria for Ax-SpA, and must be naïve of biologic therapy (anti-TNF-α agents) at the time of inclusion, or have received but subsequently discontinued anti-TNF-α therapy at least 3 months before inclusion. A blood sample will be drawn (35 mL) to these patients.
  Interventions: Other: Blood sample
- Control group (Other): Subjects must be free from any inflammatory or auto-immune disease. A blood sample will be drawn (35 mL) to these controls subjects.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — 35 mL, 7 tubes

SUMMARY:
The aim of this project is to quantify global DNA methylation in patients with Ankylosing Spondylitis or Axial Spondyloarthritis as compared with control subjects.

DETAILED DESCRIPTION:
Spondyloarthritis covers a group of diseases with common clinical, genetic and radiographic characteristics. Ankylosing spondylitis (AS) is the most common of these, and is usually diagnosed in the presence of bilateral sacroiliitis by conventional x-ray, according to the modified New York criteria. Axial spondyloarthritis (Ax-SpA) mainly affects the axial skeleton and progresses towards the formation of bone or bony structures around the sacro-iliac joint and spine, leading to the gradual formation of a bony bridge from the sacro-iliac joint and ligamentous ossifications to the spine. Early forms of the disease do not present such modifications to the sacro-iliac joint and therefore, show no visible sacroiliitis on conventional x-ray. Thus, it is possible to classify a patient aged <45 years with inflammatory lower back pain as having Ax-SpA, irrespective of the presence of sacroiliitis by x-ray. Indeed, inflammation of the sacro-iliac joint and spine occurs before the process of ossification and inflammation, and can be detected by MRI. This led the Assessment of SpondyloArthritis international Society (ASAS) group to propose candidate classification criteria for Ax-SpA, notably adapted to early forms of the disease. Accordingly, patients with Ax-SpA without radiographic sacroiliitis are considered to have non-radiographic Ax-SpA. Classification criteria for peripheral SpA are also available.

The determinants of AS and SpA are complex, and involve both genetic and environmental factors. In addition to these factors, several studies in recent years have also highlighted the emerging role of epigenetics in the pathophysiology of inflammatory diseases.

The term epigenetics refers to heritable and reversible modifications in gene expression without any change in the coding DNA sequence. This process may be involved in the pathophysiology of different diseases and their clinical expression. Several different epigenetic mechanisms may concur to modify gene functioning. Changes to the chromatin and to DNA (without modification of the encoding sequence itself) have been shown to be important for the control of gene expression through suppressive or permissive factors. Thus, DNA methylation could play a role in auto-immune or inflammatory diseases by regulating gene expression, particularly those coding for pro-inflammatory mediators such as certain cytokines, thereby contributing to dysregulation of the immune system.

DNA methylation is regulated by the activity of DNA methyltransferase enzymes (DNMT). In multicellular eukaryotic organisms, DNA methylation is associated with chromatin repression, and thereby, inhibition of gene expression. DNA methylation can be evaluated across the whole genome, but also at the level of a specific candidate gene, such as the gene encoding a pro-inflammatory cytokine.

The level of DNA methylation has been evaluated in rheumatoid arthritis (RA) and in systemic lupus erythematosus (SLE), and a "methylated-DNA" signature has been observed in these auto-immune diseases. Currently, there is no available data regarding DNA methylation in AS or SpA in general. In this study, the investigators aim to analyse the global DNA methylation in patients with AS or Ax-SpA.

ELIGIBILITY:
Inclusion Criteria:

Subjects included in the Patient group must meet the modified New York criteria for AS, or the ASAS criteria for Ax-SpA, and must be naïve of biologic therapy (anti-TNF-α agents) at the time of inclusion, or have received but subsequently discontinued anti-TNF-α therapy at least 3 months before inclusion.

Subjects included in the Control group must be free from any inflammatory or auto-immune disease. Subjects being followed for spinal disc disease (herniated disc) or abarticular mechanical disease (tendonitis) will be eligible, as well as healthy subjects.

The following inclusion criteria are common to both control and patient groups:

* Adult patients (≥18 years).
* Provide written informed consent indicating that the subject has understood the aims of the study, as well as the procedures involved, and that he/she accepts to participate and adhere to the demands and restrictions imposed by the study participation.
* All subjects must have social security coverage.
* Maximum age is 80 years.

Exclusion Criteria:

* Subjects being treated by systemic corticosteroids with a prednisone equivalent dose >10 mg/day.
* Subjects with limited legal capacity.
* Subjects judged by the investigator to be unlikely to comply with study procedures
* Subjects with no social security coverage.
* Pregnant women.
* Subjects still in the exclusion period of another study, or according to the national registry of clinical trial participants.
* Inability to understand the study objectives; psychiatric disorders deemed by the investigator to be incompatible with inclusion in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Overall level of DNA methylation | D0 (day of inclusion)
  The level of methylation will be evaluated using the global quantification technique for DNA

SECONDARY OUTCOMES:
Expression of DNMT1 and MBD2 | D0 (day of inclusion)
  Expression of DNMT1 and MBD2 will be quantified on RNA extracted from monocytes and CD4 T cells, by quantitative real-time polymerase chain reaction
Methylation of the promoter region of TNF | D0 (day of inclusion)
  Methylation of the promoter region of TNF will be evaluated on DNA from monocytes and CD4 T cells (bisulfite genomic sequencing)
Serum TNF-α | D0 (day of inclusion)
  Serum TNF-α will be quantified by ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Besançon, France

IPD SHARING:
Plan to Share IPD: No